CLINICAL TRIAL: NCT04310969
Title: Clinical Effect of MiboFlo in Dry Eye Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRECKY2019-099
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Dry Eye Syndromes; Meibomian Gland Dysfunction
Keywords: dry eye; meibomian gland dysfunction; therapy
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- treatment group (Experimental): Patients are treated every two weeks for a total of three times. Forceful expression of the meibomian glands is followed after each therapy.
  Interventions: Device: MiBoFlo Thermoflo; Procedure: forceful expression of the meibomian glands
- control group (Sham Comparator): Forceful expression of the meibomian glands only for patients.
  Interventions: Procedure: forceful expression of the meibomian glands
- active control group (Active Comparator): LipiFlow® treatment is used as an active comparator.
  Interventions: Device: LipiFlow

INTERVENTIONS:
Device: MiBoFlo Thermoflo — Each treatment for each eye takes 10 minutes and is treated every two weeks for a total of three times. The device was preheated to 42.2℃ and the eyelid was cleaned and smeared with a small amount of ultrasound gel in order to reduce friction between the device and eyelid skin. Then massage the outer skin of the upper and lower eyelids for a period of 10 minutes. The patient's eyes keep closed during therapy.
  Arms: treatment group
Procedure: forceful expression of the meibomian glands — Utilize a cotton swab on the inner surface of the eyelid and the another cotton swab on the outer lid to apply force
  Arms: control group; treatment group
Device: LipiFlow — LipiFlow treatment applies heat to the palpebral surface of eyelids while simultaneously applying graded pulsatile pressure to the outer eyelid surfaces, thereby expressing the meibomian glands during heating.
  Arms: active control group

SUMMARY:
The aim of this prospective study is to compare the changes between the patients receiving traditional treatment and the patients with MiBoFlo, evaluating the effectiveness of MiBoFlo.

DETAILED DESCRIPTION:
The MiBoFlo Thermoflo uses a proprietary thermoelectric heat pump to help meibum maximize liquefaction, improving the preservation and function of the tear film's evaporative component. It supplies continuous controlled heat to the outer skin of the eyelids, absorbing deep into the tissue and breaks down the hardened oils in the meibomian glands. We are trying to find a effective, safe and economical therapy for dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age of older;
* Meet the diagnostic criteria for dry eye developed by DEWS II: OSDI score≥15 points, TBUT≤10 minutes;
* Meet the signs of meibomian gland dysfunction

Exclusion Criteria:

* Had skin allergies or inflammation;
* Had active ocular infection or inflammation;
* Had history of ocular surgery, eyelid surgery or neurological paralysis within 6 months;
* Had history of systemic disease affecting ocular surface function, such as Stevens-Johnson syndrome, Sjögren syndrome etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
subjective symptom score | 2 weeks
  Ocular Surface Disease Index (OSDI©) questionnaire was chosen to assess subjective symptoms of dry eye, which can demonstrate sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease.
Meibomian Glands Yielding Liquid Secretion (MGYLS) | 2 weeks
  The total number of MGYLS was counted for both upper and lower lid of each eye.
Meibomian Glands Secretion (MGS) | 2 weeks
  The total number of MGYLS was counted for both upper and lower lid of each eye.

SECONDARY OUTCOMES:
Corneal Fluorescein Staining(CFS) | 2 weeks
  Fluorescein was applied in the lower conjunctival sac of each eye with a fluorescein sodium ophthalmic strip (Jingming New Technological Development Co., Ltd, Tianjin, China), and corneal erosion assessed by CFS was scored using the following grading system: grade 0 indicated no corneal erosion, grade 1 indicated 1-5 punctate epithelial erosions seen inferiorly, grade 2 indicated 6-30 punctate epithelial erosions, grade 3 indicated more than 30 punctate epithelial erosions
Tear Meniscus Height(TMH) | 2 weeks
  The lower eyelid tear meniscus was photographed under a white light source by Oculus Keratograph 5M, and TMH was measured with the built-in ruler in order to estimate tear secretion.
Non-invasive Keratograph Break-up Time(NIKBUT) | 2 weeks
  The NIKBUT was used to evaluate tear film stability and assessed by Oculus Keratograph 5M. The average NIKBUT was recorded into the statistical result.
Meibography | 2 weeks
  Meibography was performed using Meibo-Scan attached to the Oculus Keratograph 5M. Structural changes of meibomian were observed with infrared light source. Partial or complete loss of the meibomian glands was scored using the following grading system: grade 0 indicated no loss of meibomian glands, grade 1 indicated lost area less than one third of the total area of meibomian glands, grade 2 indicated lost area between one third and two thirds of total area, grade 3 indicated lost area more than two thirds of the total area

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jie, M.D, Study Director — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China